CLINICAL TRIAL: NCT05996510
Title: Investigation of the Relationship Between Suprascapular Notch Cross-sectional Area Measured by Ultrasonography and Disease Activity in Subacromial Impingement Syndrome
Brief Title: Suprascapular Notch Cross-sectional Area Measured by Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BursaYIEAH
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diseased shoulder (Active Comparator)
  Interventions: Device: ultrasound
- sturdy shoulder (Active Comparator)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Shoulder ultrasound is performed using a linear ultrasound probe. The area under the suprascapular notch and the superior transverse scapular ligament is measured using the cross-sectional area measurement method.
  Other Names: shoulder ultrasound

SUMMARY:
Chronic shoulder pain is one of the most common diseases affecting the quality of life today. Although there are multiple causes, one of the most common causes is shoulder impingement syndrome.

Ultrasound can be used for diagnosis in patients whose treatment is difficult due to its complex structure. While the supraspinatus muscle, tendon and shoulder joint are the regions that are usually evaluated, the visualization of the Suprascapular notch is usually observed during injection. The connection between the suprascapular notch and the shoulder joint has been demonstrated in different studies.

DETAILED DESCRIPTION:
In this study, the investigation of the relationship between the measurements of the suprascapular nerve and the suprascapular notch, which the investigators observed in our clinical ultrasound applications, and the disease activity intended.

ELIGIBILITY:
Inclusion Criteria:

* chronic shoulder pain
* 35-65 years
* who agreed to participate in the study

Exclusion Criteria:

* . Lymphoproliferative diseases and other neoplasms
* .Uncontrolled arterial hypertension
* Metabolic syndrome
* Uncontrolled diabetes mellitus
* Mental retardation
* Antidepressant use
* Autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Suprascapular notch cross-sectional area measurement | baseline
  The area under the suprascapular notch and the superior transverse scapular ligament is measured using the cross-sectional area measurement method.

SECONDARY OUTCOMES:
Visual Analogue Scale | baseline
  Visual Analog Scale was used for pain. Pain intensity was measured using 0-10 cm visual analogue scale (VAS). The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
Shoulder Pain and Disability Index (SPADI) | baseline
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with activity of daily livings requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items.To score either version of the SPADI, the total score is calculated by averaging the pain and disability subscale scores to find a score out of 100. On this scale, 0 represents less disability while 100 represents greatest disability

CONTACTS AND LOCATIONS:
Overall Officials: korgün ökmen, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Lale altan inceoğlu, phd, Study Chair — uludağ university faculty of medicine; ugur ertem, M.D., Study Chair — uludağ university faculty of medicine
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No